CLINICAL TRIAL: NCT06373185
Title: Comparison of the Effects of Sacral Erector Spinae Plane Block and Caudal Block on Postoperative Pain Control in Pediatric Urogenital Surgery Cases
Brief Title: Comparison of the Efficacy of Sacral Espb and Caudal Block for Pain Management After Urogenital Surgeries in Children
Acronym: SESPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Bilge Olgun Keles, Assistant Professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/21
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Urogenital Diseases; Nerve Block; Pain, Postoperative
Keywords: sacral erector spinae plane block; caudal block; nerve block; anesthesia, general; urogenital surgery
MeSH Terms: conditions — Urogenital Diseases; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized controlled double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomisation using a closed envelope method based on computer-generated random numbers was to assign patients to two equal groups. Group 1 received midline US-guided sacral erector spinae plane block and Group 2 received caudal block. The experienced anesthetist who opened the envelope performed the block according to the group code and patients were followed postoperatively by an anesthetist blinded to which block was performed. Patients were also blinded as to which block was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SESPB (Experimental): Participants received ultrasound-guided SESPB before the surgery
  Interventions: Procedure: Ultrasound-guided sacral erector spinae plane block
- CAUDAL (Active Comparator): Participants received ultrasound-guided caudal block before the surgery
  Interventions: Procedure: Ultrasound-guided caudal block

INTERVENTIONS:
Procedure: Ultrasound-guided sacral erector spinae plane block — Patients were received ultrasound-guided sacral erector spinae plane block, 1ml/kg %0.25 bupivacaine (max 20 ml), for postoperative pain management
  Arms: SESPB
Procedure: Ultrasound-guided caudal block — Patients were received ultrasound-guided caudal block, 1ml/kg %0.25 bupivacaine (max 20 ml), for postoperative pain management
  Arms: CAUDAL

SUMMARY:
The aim of this study was to compare the efficacy of caudal block and sacral espb used as a postoperative analgesia method in urogenital pediatric surgery cases.

DETAILED DESCRIPTION:
The parents of the patients who will undergo urogenital surgery will be included in the study after being informed and written consent is obtained. They will be randomised and divided into two groups. After general anaesthesia, sacral espb will be performed in the 1st group and caudal block will be performed in the 2nd group and postoperative pain will be evaluated with Face, Leg, Activity, Cry, Consolability (FLACC) score.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-7 years undergoing paediatric urogenital surgery
* Patients in American Society of Anesthesiologist (ASA) class I-II

Exclusion Criteria:

* Patients whose parents do not give consent
* Patients with anatomical changes in the sacral region, previous surgery, scar and infection,
* Patients with known local anaesthetic allergy
* Patients for whom regional anaesthesia is contraindicated
* Known neurological or muscular disease

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Face, Leg, Activity, Cry, Consolability (FLACC) score | baseline ,and 24 hours
  The FLACC is an observational pain scale. It is widely used in the paediatric population to assess pain in infants and children who are unable to verbally express their pain.Each category is scored on the 0-2 scale which results in a total score of 0-10.

SECONDARY OUTCOMES:
Analgesic requirement | baseline, and 24 hours
  If the FLACC>4 and above rescue analgesics will be made
Satisfaction of the patient's parents | 24. hours
  A questionnaire will be used in which patient's parents will indicate their satisfaction from 0 to 10. 0: not at all satisfied, 10: very satisfied
Satisfaction of the surgeons | 24.hours
  A questionnaire will be used in which surgeon's will indicate their satisfaction from 0 to 10. 0: not at all satisfied, 10: very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Olgun Keleş, Principal Investigator — Giresun University; Dilek Yeniay, Study Chair — Giresun University; Elvan Tekir Yılmaz, Study Chair — Giresun University; İlke Tamdoğan, Study Chair — Giresun University; Mehmet Değermenci, Study Chair — Giresun University
Locations (1):
- Giresun Research and Training Hospital, Giresun, Central, Turkey (Türkiye)